CLINICAL TRIAL: NCT07177937
Title: An Open-Label, Multicenter, First-in-Human, Dose-Escalation and Expansion Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of DXC014 for Injection in Patients With Advanced Solid Tumors.
Brief Title: A Study of DXC014 in Patients With Advanced Solid Tumors.
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou DAC Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DXC014-001
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Small Cell Lung Cancer; Melanoma; Prostate Cancer; Other Advanced Solid Tumors
MeSH Terms: conditions — Small Cell Lung Carcinoma; Melanoma; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Dose Escalation DXC014, Cohort Expansion DXC014
  Interventions: Drug: DXC014

INTERVENTIONS:
Drug: DXC014 — Dose Escalation DXC014, Cohort Expansion DXC014

SUMMARY:
This is a phase I, open-label, first-in-human clinical study designed to evaluate the safety, tolerability, MTD, DLT, RP2D, the PK characteristics, preliminary anti-tumor activity, the immunogenicity of DXC014 in patients with Advanced Solid Tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form and comply with the protocol requirements.
2. Male or female.
3. For other solid tumor patients: Age ≥18 years and ≤75 years；For prostate cancer patients: Age ≥18 years.

4 .Life expectancy ≥ 3 months. 5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.

6. Prostate cancer,other solid tumors. 7. Prostate Cancer (Two Parallel Cohorts): Cohort 1: At least one measurable lesion as defined by RECIST v1.1. Cohort 2: Presence of ≥1 metastatic lesion(s) confirmed by baseline CT, MRI, or bone scan.Participants and their partners agree to use effective methods of contraception (excluding the rhythm method) from the time of signing the informed consent form until 6 months after the last dose of study drug.

Other Solid Tumors: At least one measurable lesion as defined by RECIST v1.1. 8. Toxicities from prior anti-tumor therapy have recovered to Grade ≤1 as defined by NCI-CTCAE v5.0 (except alopecia). Grade 2 toxicities per NCI-CTCAE v5.0 may be permitted if judged by the investigator to pose no safety risk.

9. Adequate organ function as defined by the following laboratory values: Hematological:(1) Absolute Neutrophil Count (ANC) ≥ 1.5 × 10⁹/L (No use of G-CSF or granulocyte-/white blood cell-boosting drugs within 7 days prior to the screening lab test). (2) Platelet count ≥ 100 × 10⁹/L (No platelet or whole blood transfusion or platelet-boosting drugs within 7 days prior to the screening lab test). (3) Hemoglobin (HGB) ≥ 90 g/L (No red blood cell (RBC) or whole blood transfusion or hemoglobin-boosting drugs within 7 days prior to the screening lab test).Hepatic: (1) Total Bilirubin (TBIL) ≤ 1.5 × ULN (Upper Limit of Normal); except for participants with congenital bilirubinemia, e.g., Gilbert's syndrome (Direct bilirubin ≤ 1.5 × ULN). (2) AST and ALT ≤ 3.0 × ULN. (3) AST and ALT ≤ 5.0 × ULN in the presence of liver metastases. Renal: Creatinine Clearance (Ccr) ≥ 60 mL/min OR Serum Creatinine (Cr) ≤ 1.5 × ULN. For participants with urinalysis showing urine protein ≥ 2+ at screening, a 24-hour urine protein quantification should be performed; participants with a 24-hour urine protein ≤ 1 g may be enrolled. Coagulation: (1) International Normalized Ratio (INR) ≤ 1.5. (2) Activated Partial Thromboplastin Time (APTT) or Prothrombin Time (PT) ≤ 1.5 × ULN. Cardiac: Left Ventricular Ejection Fraction (LVEF) ≥ 50%.

10. Participants and their partners agree to use effective methods of contraception (excluding the rhythm method) from the time of signing the informed consent form until 6 months after the last dose of study drug.

Exclusion Criteria:

1. Within 14 days prior to the first dose: Underwent plasmapheresis; received systemic corticosteroid therapy at a dose >10 mg/day prednisone or equivalent for more than 3 consecutive days, or other anti-inflammatory drugs with equivalent activity (short-term use for preventing contrast agent allergy is allowed for enrollment).
2. Received systemic anti-tumor therapy or investigational drug treatment within 28 days or 5 half-lives (whichever is shorter) prior to the first dose; received palliative radiotherapy within 14 days prior to the first dose; received treatment with Chinese patent medicines or herbal medicines explicitly indicated for anti-tumor purposes in the NMPA-approved drug label within 1 week prior to the first dose.
3. History of solid organ transplantation.
4. Prostate Cancer: Leptomeningeal metastasis or brain metastasis. Other Solid Tumors: Participants with active central nervous system (CNS) metastases and/or leptomeningeal metastases or spinal cord compression, with the following exceptions: asymptomatic and stable brain metastases, or participants who have received treatment for brain metastases with no evidence of new or enlarging brain metastases on imaging for at least 4 weeks and no related symptoms, and who have discontinued steroid or anticonvulsant therapy for at least 14 days prior to initiation of study treatment.
5. Evidence of cardiovascular risk, including any of the following: a. QTcF interval ≥ 470 milliseconds (QT interval must be corrected using Fridericia's formula [QTcF]). b. Evidence of current clinically significant untreated arrhythmias, including clinically significant ECG abnormalities such as 2nd-degree (Mobitz Type II) or 3rd-degree atrioventricular block. c. History of myocardial infarction, acute coronary syndrome (including unstable angina), coronary angioplasty, stenting, or bypass grafting within 6 months prior to screening. d. Class III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system. e. Uncontrolled severe hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg).
6. Uncontrolled diabetes mellitus.
7. Current interstitial lung disease or pulmonary fibrosis, pneumoconiosis, radiation pneumonitis, severely impaired pulmonary function, or other conditions that may interfere with the detection or management of suspected drug-related pulmonary toxicity.
8. History of or current other malignancies within the past 5 years. Participants may be enrolled in the following two scenarios: other malignancies treated with single surgery alone, achieving continuous 5-year disease-free survival (DFS); adequately treated carcinoma in situ with no evidence of recurrence, such as cervical carcinoma in situ, non-melanoma skin cancer, and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ), and T1 (tumor infiltrating basement membrane)].
9. Presence of severe unhealed wounds, ulcers, or fractures; major surgery within 28 days prior to the first dose or anticipated major surgery during the clinical study period.
10. History of allergy to any component or excipient of DXC014 .
11. Active hepatitis B (HBsAg positive and HBV DNA ≥ 500 IU/mL or above the upper limit of normal [ULN] of the testing unit); active hepatitis C (HCV antibody positive and HCV RNA above the lower limit of detection).
12. Known positive HIV serology; active syphilis (participants with only a positive syphilis antibody test may be enrolled); suspected active tuberculosis (chest imaging within 3 months prior to the first dose suggests active tuberculosis infection).
13. Active bleeding within 30 days prior to screening, or judged by the investigator to be at risk of major gastrointestinal bleeding, hemoptysis, etc.; or hereditary bleeding tendency or coagulation dysfunction; or hemorrhagic symptoms requiring other medical intervention.
14. History of severe arterial/venous thrombotic events within 6 months prior to the first dose, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis, pulmonary embolism.
15. Female participants who are pregnant (positive serum pregnancy test) or breastfeeding.
16. Active infection requiring systemic medication (CTCAE ≥ Grade 2) within 2 weeks prior to the first dose of study treatment; uncontrolled pleural effusion, ascites, or pericardial effusion requiring repeated drainage.
17. Administration of a live attenuated vaccine within 28 days prior to the first dose or planned vaccination during the study period.
18. Any other condition that, in the judgment of the investigator or sponsor, may affect the participant's participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-10-20 (Estimated); Primary Completion 2030-10-20 (Estimated); Study Completion 2030-10-20 (Estimated)

PRIMARY OUTCOMES:
Number of participants that experienced dose limiting toxicities(DLTs) at given dose level. | 28 days
  Dose Limiting Toxicities (DLTs) In Order to Determine the Maximum Tolerated.
Number of participants with adverse events (AEs) | After first infusion of study drug, Through study completion an average of 1 year
  The adverse events will be evaluated in accordance with CTCAE v5.0. The investigator shall assess the relationship between the events and investigational product.

SECONDARY OUTCOMES:
Maximum observed serum or plasma concentration (Cmax) | Through study completion an average of 1 year
  One of the pharmacokinetics parameters for DXC014 investigator shall assess the relationship between the events and investigational product.
Maximum serum drug time（Tmax） | Through study completion an average of 1 year
  One of the pharmacokinetics parameters for DXC014

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Hunan Cancer Hospital, Changsha, Hunan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No